CLINICAL TRIAL: NCT06757244
Title: DOVIPA, a Phase II Study Evaluating Efficacy and Safety of DOstarlimab and Oral VItamin D3 With Folinic Acid, 5FU, Irinotecan Plus Oxalipaltin (mFOLFIRINOX) in Non Pretreated Metastatic PAncreatic Cancer
Brief Title: DOVIPA, a Study Evaluating Efficacy and Safety of DOstarlimab and VItamin D3 With mFOLFIRINOX in PAncreatic Cancer
Acronym: DOVIPA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hopital Foch (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023_0111; 2023-510004-49-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-27; First posted 2025-01-03 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Pancreas Neoplasms
Keywords: Pancreatic adenocarcinoma; metastatic PAncreatic Cancer; dostarlimab; vitamin D3; mFolfirinox; LV5FU
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — dostarlimab; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Methodology: prospective, multicentric, non-randomised, open-label, safety-run in, phase 2 study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination of mFOLFIRINOX plus dostarlimab and oral vitamin D3 (Experimental): Patients will be included and treated according to the following treatment regimen:
  * Intra-venous (i.v) dostarlimab: day1 - d21: 500mg IV q3Weeks (cycle 1 to cycle 4) then 1000 mg IV q6Weeks (from cycle 5 onwards)
  * Oral vitamin D3 8000 IU/d for 14 days, then 4000IU/d
  * mFOLFIRINOX d1, d15, d29 is administered as follow: oxaliplatin 85 mg/m2 on day1, IV infusion over 2 h, immediately followed by folinic acid 400 mg/m2 or calcium levofolinate 200 mg/m2 given as a 2-h IV infusion, with the addition of irinotecan 180 mg/m2 as per dose-level given as a 90-min intravenous infusion through a Y-connector immediately followed by 5- fluorouracil 2400 mg/m2 over 46 h continuous infusion (cycle 1 to cycle 4). From cycle 5, the mFolfirinox will be substituted by LV5FU D1, D15 and D29.
  Interventions: Drug: Dostarlimab; Drug: Vitamin D3 (Cholecalciferol); Drug: mFOLFIRINOX Treatment Regimen; Drug: LV5FU2

INTERVENTIONS:
Drug: Dostarlimab — Intra-venous (i.v) dostarlimab: day1 - d21: 500mg IV q3Weeks (cycle 1 to cycle 4) then 1000 mg IV q6Weeks (from cycle 5 onwards)
Drug: Vitamin D3 (Cholecalciferol) — Oral vitamin D3 8000 IU/d for 14 days, then 4000IU/d
Drug: mFOLFIRINOX Treatment Regimen — mFOLFIRINOX d1, d15, d29 cycle 1 to cycle 4 is administered as follow: oxaliplatin 85 mg/m2 on day1, IV infusion over 2 h, immediately followed by folinic acid 400 mg/m2 or calcium levofolinate 200 mg/m2 given as a 2-h IV infusion, with the addition of irinotecan 180 mg/m2 as per dose-level given as a 90-min intravenous infusion through a Y-connector immediately followed by 5- fluorouracil 2400 mg/m2 over 46 h continuous infusion.
Drug: LV5FU2 — folinic acid 400 mg/m2 Or calcium levofolinate 200 mg/m2 2-h IV infusion 5- fluoro-uracil 2400 mg/m2 Over 46 h continuous infusion. From cycle 5 onwards, D1=D43

SUMMARY:
The goal of this clinical trial is to estimate the antitumor response of mFOLFIRINOX + Dostarlimab + oral HD vitamin D3 in patients with non-pretreated histologically confirmed metastatic Stage IV adenocarcinoma of the pancreas. The patients must have an Eastern Cooperative Oncology Group (ECOG)-Performance Status (PS) 0 or 1 and adequate organ functions.

The main objective of the study will be assessed by estimating Objective response rate (ORR) according to Response Evaluation Criteria version 1.1 (RECIST 1.1) in patients with pancreatic adenocarcinoma and measurable disease.

The Secondary objectives are :

* To assess the safety and tolerability of mFOLFIRINOX + Dostarlimab + HD Vitamin D according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 by evaluating the Median Progression Free Survival (mPFS) in months, the Median Overall Survival (mOS) in months, the Median Duration of Response (mDOR) in months and Clinical benefit rate according to RECIST 1.1 (CBR)
* To further evaluate the antitumor efficacy of mFOLFIRINOX + Dostarlimab + oral HD Vitamin D by evaluating the type, frequency, and severity of treatment-emergent adverse events (TEAEs); adverse events of special interest (AESIs); safety laboratory findings There are also exploratory objectives to better understand the pancreatic adenocarcinoma.

Participants will be cared for in the digestive oncology department. A selection review will be carried out to check compliance with the study eligibility criteria. Patients included in the study will be treated with 4 cycles of induction therapy. Each cycle lasts 6weeks and includes chemotherapy such as mFolfirinox D1,D15 and D29, combined with dostarlimab 500 mg every 3 weeks and daily oral vitamin D3.

At the end of the induction treatment period, maintenance treatment will be instituted with LV5FU chemotherapy combined with dostarlimab 1000 mg every 6 weeks and daily oral vitamine D3. Treatment will be maintained until progression or unacceptable toxicity.

Throughout this period, patients will be monitored for their safety. Imaging examinations will also be carried out to monitor the progression of tumour disease.

ELIGIBILITY:
Inclusion criteria

1. Histologically confirmed metastatic Stage IV adenocarcinoma of the pancreas
2. No prior treatment for stage IV pancreatic adenocarcinoma (prior adjuvant or neoadjuvant treatment is not allowed)
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1
4. Male and female patients 18 - 75 years
5. Measurable disease determined using guidelines of Response Evaluation Criteria In Solid Tumors (RECIST version 1.1)
6. Accessible tumor tissue available for fresh biopsy
7. Expected survival >3 months
8. Men and women of child-bearing potential must agree to use adequate contraception.

   A female participant is eligible to participate if she is not pregnant or breastfeeding and at least one of the following conditions applies:
   * Is not a woman of childbearing potential (WOCBP), or
   * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), from the screening visit to at least 6 months after the last dose of study treatment, and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of dostarlimab, and A WOCBP must have a negative highly sensitive pregnancy test (urine or serum, as required by local regulations) within 72 hours before the first dose of study treatment.

   Fertile men who are sexually active with a WOCBP must use a male condom plus spermicide during the trial and for 6 months after the last dose of study treatment administration. Male patients should also refrain from sperm donation throughout this period.
9. Laboratory values ≤1 week prior to randomization must be Adequate hematologic values

   * Platelet count ≥100,000 cells/mm3
   * Absolute neutrophil count [ANC] ≥1,500 cells/mm3
   * Hemoglobin ≥9 g/dL or ≥90 g/L) Adequate hepatic function
   * Aspartate aminotransferase [AST/SGOT] ≤2.5x Upper Normal Limit [UNL] (≤5x UNL if liver metastases present)
   * Alanine aminotransferase [ALT/SGPT] ≤ 2.5x Upper Normal Limit (≤5x UNL if liver metastases present)
   * Bilirubin ≤1.5x UNL
   * Serum albumin > 3.0 g/dL Adequate renal function serum creatinine clearance CLcr ≥ 50 mL/min) (Cocroft-Gault Formula should be used for CrCl calculation) For participants not taking warfarin: INR <1.5 or PT <1.5 x ULN and either PTT or aPTT <1.5 x ULN. Participants taking warfarin may be included on a stable dose with a therapeutic INR <3.5 Uracilemia < 16 ng/ml
10. Patients with history of hepatitis C (HCV) infection are eligible if HCV viral load is undetectable at screening. HCV screening tests are not required unless there is a known history of HCV infection.
11. No evidence of active infection and no serious infection within the past 30 days.
12. Patient able to understand and willing to sign and date the written voluntary informed consent form at screening visit prior to any protocol-specific procedures
13. Patient affiliated to a social security regimen

Non-inclusion criteria

1. Endocrine or acinar pancreatic carcinoma
2. Participant has cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal/gastric varices, or persistent jaundice.

   Note: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) is acceptable if participant otherwise meets entry criteria.
3. Major surgical procedure, significant traumatic injury within 28 days prior to study treatment start. Incompletely healed wounds or anticipation of the need for major surgical procedure during the course of the study
4. Known cerebral metastases, central nervous system (CNS), or epidural tumor
5. Prior anticancer treatment for adenocarcinoma of the pancreas including prior adjuvant or neoadjuvant treatment
6. Known dose tivity reaction to any of the components of study treatments.
7. Pregnancy (absence to be confirmed by β-hCG test) or breast-feeding period
8. Clinically relevant coronary artery disease or history of myocardial infarction in the last 6 months, or high risk of uncontrolled arrhythmia (for men: QTc ≥450 msec, for women: QTc ≥470 msec). Inclusion of patients with hypokalemia, hypomagnesemia and hypocalcemia (defined as results less than normal in Baseline testing) is not allowed.
9. Previous malignancy in the last 5 years except curative treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix
10. History or current evidence on physical examination of central nervous system disease or peripheral neuropathy ≥ grade 1 Common Toxicity Criteria for Adverse Events (CTCAE) v5.0.
11. Any significant disease which, in the investigator's opinion, would exclude the patient from the study.
12. Patient with a DPD deficiency or UGT1A1 homozygous 7/7; the test should be done for all patients before 5-FU administration, according to ANSM communication regarding recommendation about high risk of no testing DPD in patient before 5-FU administration
13. Has undergone prior allogeneic hematopoietic stem cell transplantation
14. Has had an allogeneic tissue/solid organ transplant
15. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent)
16. Participant has received systemic steroid therapy (>10 mg daily prednisone or equivalent) within 7 days before the first dose of the study treatment or is receiving any other form of immunosuppressive medication. Replacement therapy (adrenal or pituitary insufficiency) is not considered a form of systemic therapy. Use of inhaled corticosteroids, local steroid injection, or steroid eye drops is allowed.
17. Participant has received a live vaccine within 30 days of planned start of study therapy. COVID-19 vaccines that do not contain live viruses are allowed. Note: mRNA and adenoviral-based COVID-19 vaccines are considered non-live.
18. History of or serology positive for HIV
19. Patients who have documented presence of HBsAg [or HBcAb] at Screening or within 3 months prior to first dose of study intervention are excluded. HBV screening tests are not required unless there is a known history of HBV infection.
20. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
21. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
22. Has an active infection requiring systemic therapy
23. Allergy: Participant cannot have history of severe allergic and/or anaphylactic reactions to chimeric, human or humanized antibodies or fusion proteins, sensitivity to any of the study treatments or components thereof, or a history of drug or other allergy that contraindicates their participation.

    In accordance with the updated SmPC of the products used in this trial, patient cannot be included in the following conditions:
    * patient has a peripheral sensitive neuropathy with functional impairment prior to first course (contra-indication use with Oxaliplatin)
    * concomitant use with St John's Wort - Chronic inflammatory bowel disease and/or bowel obstruction (contra-indication with Irinotecan)
    * patient which has been treated with brivudine, sorivudine or their chemically related analogues, which are potent inhibitors of the enzyme dihydropyrimidine dehydrogenase (DPD), which degrades fluorouracil. Fluorouracil must not be taken within 4 weeks of treatment with brivudine, sorivudine or their chemically related analogues (contra-indication with fluorouracil)
    * patient has diseases/conditions associated hypercalcaemia and / or hypercalciuria. - Calcium nephrolithiasis, nephrocalcinosis, D- hypervitaminosis
24. Being deprived of liberty or under guardianship
25. Potential participants who are pregnant, breastfeeding, or expecting to conceive children while receiving study treatment and/or unwilling to use highly effective contraception for up to 6 months after the last dose of study treatment are not eligible for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2028-02-18 (Estimated); Study Completion 2028-02-18 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) according to Response Evaluation Criteria version 1.1 (RECIST 1.1) in patients with pancreatic adenocarcinoma and measurable disease | 24 months
  The proportion of patients with an objective response at the completion of their follow-up (truncated at 24 months), among all eligible patients. An objective response will be defined as the best overall response of complete response (CR) or partial response (PR) assessed by investigators using validated criteria (i.e. RECIST 1.1)

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) as assessed by CTCAE v5.0. | From the initiation of study treatment until 90 days after the last dose or 30 days following cessation of study intervention if the participant initiates new anticancer therapy, whichever is earlier, assessed up to 24 months"
  The number and percentage of participants experiencing at least one treatment-emergent adverse event (TEAE) will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. TEAEs are defined as adverse events occurring after the initiation of study treatment and before 90 days after the last dose or 30 days following cessation of study intervention if the participant initiates new anticancer therapy, whichever is earlier, must be reported by the investigator, or an already present event that worsens in intensity or frequency following the treatment. TEAEs will be categorized by type (serious or non-serious; expected or unexpected) and severity (CTCAE grades 1 to 5) as per investigator assessment
Incidence of participants with adverse events of special interest (AESIs) as assessed by CTCAE v5.0. | From the initiation of study treatment until 90 days after the last dose or 30 days following cessation of study intervention if the participant initiates new anticancer therapy, whichever is earlier, assessed up to 24 months"
  The number and percentage of participants experiencing at least one adverse events of special interest (AESIs) will be summarized. AESIs are pre-defined events requiring detailed monitoring and rapid communication by the investigator due to their potential association with the investigational product. The severity of AESIs will be graded using CTCAE v5.0 (CTCAE grades 1 to 5).
Number of Participants With Clinically Significant Changes in Hematology, Clinical Chemistry, Thyroid Function and Urinalysis Lab Parameters | From the initiation of study treatment until 90 days after the last dose or 30 days following cessation of study intervention if the participant initiates new anticancer therapy, whichever is earlier, assessed up to 24 months"
  Blood and urine samples will be collected to evaluate hematology, clinical chemistry, thyroid function and urinalysis lab parameters . Changes from baseline to post-baseline visits will be computed. Final values and changes from baseline in continuous variables will be described et each visit. Clinically significant laboratory abnormalities (as defined by CTCAE v5.0 criteria) will also be reported.
Number of Participants With AEs Leading to Death | From the initiation of study treatment until 90 days after the last dose or 30 days following cessation of study intervention if the participant initiates new anticancer therapy, whichever is earlier, assessed up to 24 months"
  Number of participants with TEAEs leading to death will be assessed.
Median Progression Free Survival (mPFS) in months | 24 months
  The median PFS will be assessed as the time after which half of the patients are progression-free and alive.
Median Overall Survival (mOS) in months | 24 months
  The median OS will be assessed as the time after which half of the patients are alive.
Median Duration of Response (mDOR) in months | 24 months
  the time from onset of first response (PR or CR as defined above) to progression or death due to any reason, whichever occurs first
Number of Participants With Immune Related Adverse Events (irAEs) | From the initiation of study treatment until 90 days after the last dose or 30 days following cessation of study intervention if the participant initiates new anticancer therapy, whichever is earlier, assessed up to 24 months"
  The irAEs are events which may be severe or fatal according to CTCAE v5.0 and can occur in participants treated with monoclonal antibodies directed against immune checkpoints, including dostarlimab While irAEs (eg, diarrhea/colitis, pneumonitis, nephritis, hypophysitis, adrenalitis, thyroiditis, severe skin reactions, uveitis, myocarditis, and hepatotoxicity) usually occur during treatment, symptoms can also manifest after discontinuation of treatment.
Clinical benefit rate according to RECIST 1.1 (CBR) | 24 months
  the proportion of patients with the Best Overall Response equal to Complete Response, Partial Response or Stable Disease, among all eligible patients.
Number of Participants With Adverse Events Leading to Discontinuation | From the initiation of study treatment until 90 days after the last dose or 30 days following cessation of study intervention if the participant initiates new anticancer therapy, whichever is earlier, assessed up to 24 months"
  An AE is any event that was not present prior to the initiation of study treatment or any eventalready present that worsens in either intensity or frequency following exposure to study treatment. Number of participants with adverse events leading to discontinuation will be assessed.
Incidence of patient premature discontinuations (due to SAE or non-adherence to protocol) | From the initiation of study treatment until premature discontinuation due to serious adverse event or non adherence to protocol whichever is earlier, assessed up to 24 months"
  Incidence of serious adverse events or non adherence to protocol leading to discontinuation will be assessed.
Incidence of dose modifications | From the initiation of study treatment until the last dose administration, assessed up to 24 months"
  Incidence of dose modifications due to the appearance of AEs (measured in dose modification compared with the protocol planned dose of treatments)
Incidence of delays or interruptions in the administration of treatment due to the appearance of AEs | From the initiation of study treatment until the last dose administration, assessed up to 24 months"
  Incidence of delays or interruptions in the administration of treatment due to the appearance of AEs (measured in days or weeks since the initial scheduled date of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Jaafar BENNOUNA, Pr, Study Director — Hôpital Foch
Locations (5):
- France (5):
  - Marseille CRLCC, Marseille
  - CHU Hôtel Dieu, Nantes
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No
The results of study will be shared as Aggregate data results in the study publication. There is no need to share IPD.